CLINICAL TRIAL: NCT01254240
Title: Randomized Double-blind Phase 2 Study of Impact of Ultraviolet A (UVA) on Pruritus During Ultraviolet A/B (UVA/B) Phototherapy of Inflammatory Dermatoses
Brief Title: Efficacy Study of Two Choices of Phototherapy on Itching Skin Diseases
Acronym: PRUVAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DER-USZ-AAN-005
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Eczema; Psoriasis
MeSH Terms: conditions — Eczema; Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UVA/B phototherapy treatment (Experimental): UVA/B phototherapy units, stand alone cabins, patients undress, step in the cabin and receive treatment in a duration of seconds to minutes. The noticable difference between the UVA/B and UVB treatment is only in the settings of the cabin.
  Interventions: Device: UVA / UVB phototherapy
- UVB phototherapy treatment (Active Comparator): UVB phototherapy units, stand alone cabins, patients undress, step in the cabin and receive treatment in a duration of seconds to minutes. The noticable difference between the UVA/B and UVB treatment is only in the settings of the cabin.
  Interventions: Device: UVB phototherapy

INTERVENTIONS:
Device: UVA / UVB phototherapy — UVA / UVB phototherapy
  Other Names: Waldmann phototherapy cabins
  Arms: UVA/B phototherapy treatment
Device: UVB phototherapy — UVB phototherapy
  Other Names: Waldmann phototherapy cabins
  Arms: UVB phototherapy treatment

SUMMARY:
This is a double-blind prospective randomized monocenter study comparing the efficacy of two phototherapy ultraviolet spectra on pruritus (itching) of inflammatory skin diseases. 40 patients per treatment, in total 80 study participants.

DETAILED DESCRIPTION:
In patients with a skin disease and the given indication for a phototherapy with Ultraviolet B narrow-band (UVB narrowband, 311nm) with or without Ultraviolet A (UVA, 320-400 nm), the subjective pruritus levels and clinical severity will be measured before, during and after completion of the 16-week therapy (40 patients per group). Patients will be recruited in the department of dermatology of the University Hospital Zürich in the outpatient clinic. Following oral and written consent, pruritus levels will be measured by a visual analogue scale and a new, detailed pruritus score 2 before start of therapy, every 4 weeks after start as well as after completion of the phototherapy. Phototherapy is to be administered 3 times per week. The study includes 5 study visits and up to 43 treatment visits that include administration of phototherapy only.

A physical examination including clinical scores (Psoriasis Area and Severity Index PASI, Eczema Area and Severity Index EASI, Physician's static global assessment PSGA and Dermatology Dynamics Vector DDV) will be performed at every visit. During the first physical examination the Fitzpatrick-skin type of patient will be recorded, the demographics, the Body Mass Index (BMI), diagnosis, past medical history, co-morbidities, concomitant medication and the number of past UVA/B treatments.

ELIGIBILITY:
Inclusion criteria:

- Pruritic inflammatory diseases such as atopic dermatitis, other types of eczema, psoriasis, prurigo simplex subacuta and others.

Main inclusion criteria:

* Pruritus VAS Score 5 or higher at screening.
* Dermatological indication for a phototherapy with UVB nb / UVA
* Oral and written informed patient consent

Exclusion criteria:

- Patients will be excluded from the study if they fulfill any of the following criteria:

1. Foreseeable interruption of the light therapy for more than 14 days, or interruption of the light therapy for more than 14 days during the study
2. Heightened photosensitivity for UVA or UVB
3. Withdrawal of consent to participate
4. Concomitant participation in another study or having taken part in another clinical study within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
5-D Pruritus score and VAS Score at 16 weeks | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Hofbauer, MD, Leading Physician, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Zurich, Department of Dermatology, Zurich, Switzerland